CLINICAL TRIAL: NCT00804869
Title: Standard A-mode Ultrasonography vs PalmScan Ultrasonography: Biometric Measurements.
Brief Title: A-mode vs PalmScan Ultrasonography: Biometric Measurements.
Status: Withdrawn | Type: Observational
Why Stopped: Undefined
Sponsor: Asociación para Evitar la Ceguera en México (Other)
Responsible Party: Sponsor
Other Study IDs: APEC-037
Record Dates: First submitted 2008-12-03; First posted 2008-12-09 (Estimated); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Axial Length (AL); Anterior Chamber Deep (ACD); Lens Thickness (LT)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1: PalmScan biometric group
  Interventions: Device: PalmScan A2000 ultrasonography system (Micro Medical Devices, Calabasas, CA)
- 2: A-mode ultrasonography biometric group
  Interventions: Device: Standard A-mode ultrasound (Eye Cubed™, Ellex, Adelaide, Australia).

INTERVENTIONS:
Device: PalmScan A2000 ultrasonography system (Micro Medical Devices, Calabasas, CA) — PalmScan biometric measurements
  Groups: 1
Device: Standard A-mode ultrasound (Eye Cubed™, Ellex, Adelaide, Australia). — A-mode biometric measurements group
  Groups: 2

SUMMARY:
Ultrasonography has become a critical ancillary test in the clinical practice of ophthalmology. It is commonly used as a standardized method for assessing intraocular biometry. The PalmScan ultrasonography (PsU) is a portable A-scan device that uses the same principles as the standard A-scan. The aim of the study is to compare the reliability of their measurements, in order to use them indistinctively.

ELIGIBILITY:
Inclusion Criteria:

* Patients with indication for a standard A-mode ultrasound

Exclusion Criteria:

* No superficial anormalities.
* Patients with external injuries.
* Intraocular silicon oil.
* Retinal detachment
* Significant ocular pathologies.

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients who need axial length calculation.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2008-10 (Actual); Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
axial length (AL). | during examination
Anterior Chamber Deep (ACD) | during examination
Lens Thickness (LT) | during examination

CONTACTS AND LOCATIONS:
Locations (1):
- Asociación para Evitar la Ceguera en México, Mexico City, Mexico City, Mexico